CLINICAL TRIAL: NCT01319604
Title: Randomized Clinical Investigation to Assess the Efficacy of SENSIMED Triggerfish Continuous IOP Monitoring
Brief Title: SENSIMED Triggerfish
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 10/01
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Study device during 3 hours (Experimental)
  Interventions: Device: SENSIMED Triggerfish
- Study device during 6 hours (Experimental)
  Interventions: Device: SENSIMED Triggerfish
- Study device during 9 hours (Experimental)
  Interventions: Device: SENSIMED Triggerfish
- Study device during 12 hours (Experimental)
  Interventions: Device: SENSIMED Triggerfish
- Study device during 15 hours (Experimental)
  Interventions: Device: SENSIMED Triggerfish
- Study device during 18 hours (Experimental)
  Interventions: Device: SENSIMED Triggerfish
- Study device during 21 hours (Experimental)
  Interventions: Device: SENSIMED Triggerfish
- Study device during 24 hours (Experimental)
  Interventions: Device: SENSIMED Triggerfish
- Tonometric assessment during 24 hours (Active Comparator)
  Interventions: Device: Tonometer

INTERVENTIONS:
Device: SENSIMED Triggerfish — Soft contact lens-based device for the continuous monitoring of IOP fluctuations
  Arms: Study device during 12 hours; Study device during 15 hours; Study device during 18 hours; Study device during 21 hours; Study device during 24 hours; Study device during 3 hours; Study device during 6 hours; Study device during 9 hours
Device: Tonometer — Tonometric assessment of IOP
  Arms: Tonometric assessment during 24 hours

SUMMARY:
The purpose of the investigation is to investigate the relationship between the study device output and tonometric assessments.

DETAILED DESCRIPTION:
60 subjects will be enrolled in total. Enrolled patients will be randomized into one of 8 device groups of 6 subjects each or into the control group containing 12 subjects. Patients in the device arm will receive one session of 3-to 24-hour continuous IOP monitoring with SENSIMED Triggerfish®. SENSIMED Triggerfish® monitoring will begin at 18h ± 2 hours for all patients. SENSIMED Triggerfish® will be installed randomly on right or left eyes. During SENSIMED Triggerfish® monitoring on one eye, GAT and/or Perkins IOP measurements will be taken in the fellow eye every 3 hours. Outside this time they will receive GAT and/or IOP measurements every 3 hours in both eyes until the end of the 24-hours period. Patients in the control group will receive GAT and/or ICare PRO IOP measurements every 3 hours for 24 hours in both eyes.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent for the investigation
* Confirmed diagnosis of primary open angle glaucoma or normal tension glaucoma of similar degree in both eyes
* Age 18-85
* Stable anti-glaucomatous therapy 4 weeks before and throughout the investigation

Exclusion Criteria:

* Patients not able to understand the character and individual consequences of the investigation
* Patients with contraindications for silicone contact lens wear
* Wear of full frame metallic glasses during SENSIMED Triggerfish® monitoring
* Diagnosis of pseudoexfoliation syndrome / pseudoexfoliative glaucoma and of pigment dispersion syndrome / pigmentary glaucoma
* Severe dry eye
* Patients who have had ocular surgery within the last 3 months
* Corneal or conjunctival abnormality or irregularity hindering correct contact lens adaptation
* Allergy to corneal anaesthesia
* Simultaneous participation in other clinical research

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Relationship between study device signal and tonometer reading | during 24 hours of study device wear

CONTACTS AND LOCATIONS:
Overall Officials: Milko Iliev, MD, Principal Investigator — University of Bern
Locations (5):
- University Hospital Leuven, Leuven, Belgium
- University Hospital Glostrup, Glostrup Municipality, Denmark
- Spain (2):
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitari i Politècnic la Fe, Valencia
- Inselspital, Bern, Switzerland